CLINICAL TRIAL: NCT02681068
Title: MicroTrans - A Multicenter Registry of Fecal Microbiota Transplantation
Acronym: MicroTrans
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Maria J.G.T. Vehreschild, PD Dr. med., University of Cologne
Other Study IDs: MicroTrans
Record Dates: First submitted 2016-02-02; First posted 2016-02-12 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Clostridium Infections
Keywords: Fecal microbiota transplantation (FMT); Clostridium difficile associated diarrhea (CDAD)
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Fecal microbiota transplantation (FMT) — Fecal microbiota transplantation (FMT) for patients with Clostridium difficile associated diarrhea

SUMMARY:
The registry collects cases of patients received fecal microbiota transplantation (FMT) due to Clostridium difficile associated diarrhea (CDAD). The main objective of this study is to analyze the safety and effectiveness of FMT. Furthermore, data analysis will be used to implement a standardization of FMT in German hospitals and improve patient outcome. Therefore, a detailed description of completions of FMT are documented on our web-based survey platform www.ClinicalSurveys.net.

DETAILED DESCRIPTION:
Concerning the documentation of patients received fecal microbiota transplantation (FMT) due to Clostridium difficile associated diarrhea (CDAD), physicians from all German hospitals performing a FMT are invited to provide prospective and retrospective information on these cases. Documentation of patient is performed by using the web-based survey platform www.ClinicalSurveys.net which was set up by researchers of the University Hospital of Cologne. This survey platform enables an optimal performance in epidemiological, observational, and interventional trials and is characterized by layered access security and frequent data backup. It has been used for numerous registry and cohort studies with approval of competent authorities and ethics boards.

The following data items are retrospectively or prospectively documented into our database, depending on if a informed consent exists or not:

* Patient characteristics (age, gender, weight, height, underlying disease)
* Indication for FMT
* Administration of antibiotics, chemotherapy, and immunosuppression prior to FMT
* Bowel movement prior to FMT
* Screening prior to FMT
* Description concerning completion of FMT
* Basic informations of the donor
* Outcome
* Prospective long term follow up (10 days, four weeks, three months, six months, and 24 months)

The following two differences of data documentation are observed:

1. Retrospective data documentation:

   Data of patients without an informed consent are documented strictly retrospectively after completion of the FMT. No pseudonymization of patient data is carried out so that no re-identification is possible.
2. Prospective data documentation:

Data of patients with an informed consent prior to FMT are documented prospectively. A pseudonymization of patient data allows a post-FMT contact (by writing or phone) to patients with respect to the 10 days, four weeks, three months, six months,and 24 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Clostridium difficile associated diarrhea

Exclusion Criteria:

* Patients < 18 years old

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent Clostridium difficile infection
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-03 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants without another Clostridium difficile infection after fecal microbiota transplantation (FMT) | 24 months after FMT
  A 24 month follow-up allows analyses of long-term effects of FMT

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 24 months after FMT
  A 24 month follow-up allows analyses of long-term effects of FMT

CONTACTS AND LOCATIONS:
Overall Officials: Maria Vehreschild, MD, Principal Investigator — University Hospital of Cologne, Department of Internal Medicine / Infectious Diseases, Cologne, Germany
Locations (1):
- University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tacke D, Wisplinghoff H, Kretzschmar A, Farowski F, Koehler P, Herweg J, Cornely OA, Vehreschild MJ. First implementation of frozen, capsulized faecal microbiota transplantation for recurrent Clostridium difficile infection into clinical practice in Europe. Clin Microbiol Infect. 2015 Nov;21(11):e82-4. doi: 10.1016/j.cmi.2015.06.027. Epub 2015 Jul 8. No abstract available. PMID 26163107
- [Derived] Bestfater C, Vehreschild MJGT, Stallmach A, Tuffers K, Erhardt A, Frank T, Gluck T, Goeser F, Sellge G, Solbach P, Eisenlohr H, Storr M; German Clinical Microbiome Study Group (GCMSG). Clinical effectiveness of bidirectional fecal microbiota transfer in the treatment of recurrent Clostridioides difficile infections. Dig Liver Dis. 2021 Jun;53(6):706-711. doi: 10.1016/j.dld.2021.02.022. Epub 2021 Mar 18. PMID 33744169
- [Derived] Hagel S, Fischer A, Ehlermann P, Frank T, Tueffers K, Sturm A, Link A, Demir M, Siebenhaar A, Storr M, Glueck T, Siegel E, Solbach P, Goeser F, Koelbel CB, Lohse A, Luebbert C, Kandzi U, Maier M, Schuerle S, Lerch MM, Tacke D, Cornely OA, Stallmach A, Vehreschild M; German Clinical Microbiome Study Group (GCMSG). Fecal Microbiota Transplant in Patients With Recurrent Clostridium Difficile Infection. Dtsch Arztebl Int. 2016 Sep 5;113(35-36):583-9. doi: 10.3238/arztebl.2016.0583. PMID 27658471